CLINICAL TRIAL: NCT06410612
Title: The Effect of Regional Anesthesia and Periarticular Injection and Versus Periarticular Injection Alone on Early Recovery After Total Knee Arthroplasty: A Prospective Randomized Trial
Brief Title: Block and Periarticular Injection Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202311211
Record Dates: First submitted 2024-03-11; First posted 2024-05-13 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Conduction

STUDY DESIGN:
Intervention Model Description: patients will be randomized into 2 groups.
Who Masked: Participant
Masking Description: patients will not know which group they are in
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Block and Periarticular injection (Active Comparator): regional anesthesia (Adductor canal block +IPACK) and Periarticular injection
  Interventions: Drug: regional anesthesia and PAI; Drug: PAI
- Periarticular injectin alone (Active Comparator): Periarticular injection alone
  Interventions: Drug: PAI

INTERVENTIONS:
Drug: regional anesthesia and PAI — this is the block portion of the study
  Other Names: adductor canal block; periarticular injection
  Arms: Block and Periarticular injection
Drug: PAI — this is the no block portion of the study
  Other Names: Periarticular injections

SUMMARY:
The purpose of the study is to compare two types of perioperative analgesic modalities, adductor canal block plus interspace between popliteal artery and capsule of the knee (IPACK) block and periarticular injection versus periarticular injection alone, to determine their relative efficacies with regard to pain relief and functional outcomes in the early postoperative period following primary total knee arthroplasty.

DETAILED DESCRIPTION:
The widespread adoption of multimodal analgesia in contemporary total knee arthroplasty (TKA) has led to improvements in perioperative pain control, expedited recovery times, and shorter hospital stays1-3. Periarticular injections (PAIs), adductor canal blocks (ACBs), and interspace between popliteal artery and capsule of the knee (IPACK) blocks are commonly utilized as part of contemporary multimodal analgesia protocols, but their relative efficacies in improving early recovery after TKA has yet to be definitively elucidated4. There are a few known potential drawbacks of ACBs and IPACKs including surgical delay due to administration timing, increased costs, and small risks associated with a regional block. Both regional anesthesia and PAI have been found to be effective alone in improving pain and opioid consumption, but there is limited data on whether there is an additive benefit of providing both treatments for patients undergoing primary TKA. Therefore, the purpose of our study is to compare the efficacy of regional anesthesia and PAI vs. PAI alone for pain management and functional recovery in the early postoperative period following TKA.

Design Prospective randomized trial

Treatment Groups All ACBs will be administered as a single shot preoperatively in the holding area on the day of surgery by the regional anesthesia team and PAIs will be administered intraoperatively by the treating orthopaedic surgeon.

Group 1: regional anesthesia (ACB + IPACK) and PAI Group 2: PAI alone

ELIGIBILITY:
Inclusion Criteria:

* Planning to undergo Unilateral primary total knee arthroplasty.
* 18 and up
* Willing to sign informed consent
* Willing to return for all follow-up visits
* Smartphone or tablet device capable of running the FocusMotion platform

Exclusion Criteria:

* BMI > 45
* Preexisting functionally limiting neurologic disorders
* Hepatic or renal insufficiency
* History of unprovoked venous thromboembolism
* Inability to complete baseline functional testing
* Chronic opioid or gabapentin and pregabalin use (chronic defined as use >5 days per week prior to the surgical procedure)
* Allergy or intolerance to trial medications
* Planned admission to a postoperative rehabilitation facility
* Planned general anesthesia
* Receiving workers compensation or disability payments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Mean Visual Analog Scale (VAS) pain score for 2 weeks postoperatively | at 2 weeks
  pain score 0-10 10 being more pain

SECONDARY OUTCOMES:
daily opioid consumption | daily up to 2 weeks postop
  opioid medications survey
daily resting Visual Analog Scale (VAS) score | daily up to 2 weeks postop
  Pain score survey 0-10, 10 being more pain
daily step count | daily up to 2 weeks postop
  step count throught fitbit
length of stay | postop day 1
  in hospital stay
complications | 14 days postop
  Number of participants with complications such as revision, infection, etc
knee range of motion | daily through app and knee brace up to 2 weeks postop
  range of motion daily through app exercises
Oxford knee score | weekly up to 2 weeks postop
  oxford knee survey through app, 0-48 scale 0 being min and 48 being max
sleep quality | daily up to 2 weeks postop
  sleep quality through app surveys and fitbit data

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Schneider, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, Creve Coeur, Missouri, United States

IPD SHARING:
Plan to Share IPD: No